CLINICAL TRIAL: NCT07075133
Title: Chrono-restricted Diet and Physical Activity as a New Preventive Strategy for Sarcopenia in Postmenopausal Women With Obesity and Type 2 Diabetes
Acronym: TIMEDIAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/23/0432; 2025-A00832-47 (Registry Identifier: ID-RCB Number)
Record Dates: First submitted 2025-06-24; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Sarcopenia; Post Menopause; Type 2 Diabetes; Circadian Clock
Keywords: Timing of eating; Timing of exercise; Muscle Function; Metabolic Health; Obesity; Menopause; women
MeSH Terms: conditions — Obesity; Sarcopenia; Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet control (no chrono restriction) + exercise performed in the morning (Experimental): Patients following a standard antidiabetic diet combined with morning exercise
  Interventions: Other: Antidiabetic diet (control); Other: Physical activity in the morning
- eTRE (chrono restriction) + exercise performed in the morning (Experimental): Patients following the eTRE program combined with physical exercise performed in the morning
  Interventions: Other: eTRE diet; Other: Physical activity in the morning
- eTRE (chrono restriction) + exercise performed in the afternoon (Experimental): Patients following the eTRE program combined with physical exercise performed in the afternoon
  Interventions: Other: eTRE diet; Other: Physical activity in the afternoon

INTERVENTIONS:
Other: Antidiabetic diet (control) — Standard antidiabetic diet
  Arms: Diet control (no chrono restriction) + exercise performed in the morning
Other: eTRE diet — eTRE for a total duration of 12 weeks. During the eTRE, volunteers will have to eat and drink (meals + snacks, medication) exclusively during an 8-hour period which will extend between 6 a.m. (flexible: or 7 a.m. or 8 a.m.) in the morning and 2 p.m. (depending on the chosen start time: or 3 p.m. or 4 p.m.), which corresponds to a fasting period of 16 hours per day
  Arms: eTRE (chrono restriction) + exercise performed in the afternoon; eTRE (chrono restriction) + exercise performed in the morning
Other: Physical activity in the morning — Physical exercise will consist of 3 weekly morning sessions that will combine aerobic and resistance exercises
  Arms: Diet control (no chrono restriction) + exercise performed in the morning; eTRE (chrono restriction) + exercise performed in the morning
Other: Physical activity in the afternoon — The physical exercise will consist of 3 weekly afternoon sessions that will combine aerobic and resistance exercises.
  Arms: eTRE (chrono restriction) + exercise performed in the afternoon

SUMMARY:
The aim of TIMEDIAB is to demonstrate that early TRE (eTRE) combined to late (afternoon) exercise will outperform eTRE combined to morning exercise on muscle function as primary endpoint, and glucose homeostasis as secondary endpoint

DETAILED DESCRIPTION:
Overweight, obesity, aging and menopause are all independent risk factors in the development of type 2 diabetes mellitus (T2DM). Older women with T2DM are at especially high risk for sarcopenia, i.e. loss of skeletal muscle mass and force, and cardiovascular diseases. The first line of T2DM treatment is based on lifestyle changes including weight loss and physical activity. One major current medical challenge is to find novel lifestyle therapies able to reduce cardiometabolic risk while perserving muscle mass in obese older individuals. As a result, intermittent fasting approaches, including time-restricted feeding/eating (TRF/TRE), have been offered as alternative dietary strategies that may have beneficial effects on weight control and T2DM. It has been recently observed that long-term TRF improve glucose homeostasis while perserving muscle mass and force in female obese mice. The purpose of TIMEDIAB is to demonstrate that early TRE (eTRE) combined to late (afternoon) exercise will outperform eTRE combined to morning exercise on various components of muscle health as primary endpoint, and blood glucose control, body composition, energy balance, cardiovascular risk, and metabolic health as secondary endpoints. This study will pave the way to larger scale randomized clinical trials investigating the long-term effects/benefits of such intervention and in other target populations.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (amenorrhea for at least 12 months, confirmed by gonadotrophins measures)
* Age range 45-70 years
* T2DM diagnosed for more than 1 year
* Subjects with T2DM treated with lifestyle control alone or associated with metformine ± DPP4 inhibitors
* Ability to sign written informed consent before any study-specific procedure
* Subject considered as reliable and capable of adhering to protocol
* Subjects with Body Mass Index (BMI)≥ 30 kg/m²
* Baseline eating period ≥ 14 h per day (as estimated by 95% eating interval)

Exclusion Criteria:

* Subjects on T2DM injectable medication or drugs able to induce hypoglycemia (glinides, sulfonylurea)
* Subjects with HbA1c > 8%
* Subjects with any of the following medical conditions:

  * Congestive cardiac failure
  * Stage 4 chronic kidney disease (i.e. eGFR < 30 ml/min/1.73 m2)
  * Liver cirrhosis or chronic liver disease
  * Any medical condition that in the opinion of the investigator could jeopardize or compromise the subject's ability to participate in the study
* Subjects with previous or present history of serious eating disorder
* Subjects not able to understand the informed consent form or fasting diary instructions
* Subjects currently participating or has participated in another study of an investigational medication or an investigational medical device within the last 30 days
* Women with menopause hormone replacement therapy

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2029-07-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in skeletal muscle function | 4 years
  Change in skeletal muscle function, assessed by 30-CTS score at inclusion (baseline) and 12 weeks after diet/exercise program; This test is used to assess lower limb strength. The score corresponds to the total number of standing positions correctly performed within the allotted 30 seconds.

SECONDARY OUTCOMES:
Change in muscle function | 4 years
  Change in muscle function assessed by various tests, such as:
  - TUG Score ( calculates the time it takes to get up from a chair without using your arms. A time <10 seconds is normal; 10>time<20 is a marker of frailty; time <20 seconds:the elderly person is at high risk of falling).
• Change in M value measured by hyperinsulinemic euglycemic clamp | 4 years
  Systemic insulin sensitivity will be assessed using a euglycemic hyperinsulinemic clamp, oral hyperglycemia, and insulin signaling pathway studies. The M value (unitless measurement) determined during the clamp will be the marker of systemic insulin sensitivity.
Change in HbA1c, during an oral glucose tolerance test | 4years
  Change in HbA1c (in percentage), during an oral glucose tolerance test
Change in fasting glucose, during an oral glucose tolerance test | 4years
  Change in fasting glucose (g/l), during an oral glucose tolerance test
Change in 2h blood glucose, during an oral glucose tolerance test | 4 years
  Change in 2h blood glucose (g/l), during an oral glucose tolerance test
Change of the insulin resistance index (HOMA-IR) | 4years
  Change of the insulin resistance index (HOMA-IR) from fasting parameters: from fasting insulin levels (mU/mL) and fasting blood glucose levels (mmol/L)
Change of the insulin sensitivity index (HOMAβ) | 4years
  Change of the insulin sensitivity index (HOMAβ) from fasting parameters: from fasting insulinemia (mU/mL) and fasting blood glucose (mmol/L)
Change in body weight (kg) | 4years
Change in body mass index (kg/m2) | 4years
Change in waist circumference (cm) | 4years
Change in waist-to-hip ratio (without unit) | 4years
Change in body composition | 4years
  Change in body composition (fat mass, lean mass, bone mass, muscle mass)
Change in blood pressure | 4years
  Change in systolic and diastolic pressure (mmHg)
Change in plasma lipid profile | 4years
  Liver and muscle lipid content will be measured by MRI.
Change in muscle function | 4 years
  Change in muscle function assessed by various tests, such as: Prehension strength: The value of the hand grip strength is measured with a dynamometer for 3 to 5 seconds by 3 measurements with each hand. The average of the 3 measurements for each hand will allow the dominant hand to be interpreted
Change in muscle function | 4 years
  Change in muscle function assessed by various tests, such as: SPPB score: Assesses physical performance and distinguishes between people with severe disability (0-4 points), moderate or frail (4-6 points), mild or pre-frail (7-9 points), and those without significant disability or independent (10-12 points).
Change in visceral fat (kg) | 4 years
Change in liver fat (kg) | 4 years
Change in muscle fat (kg) | 4 years
Change in muscle function | 4 years
  Change in muscle function assessed by various tests, such as: TUG Score ( calculates the time it takes to get up from a chair without using your arms. A time <10 seconds is normal; 10>time<20 is a marker of frailty; time <20 seconds:the elderly person is at high risk of falling).
Change in muscle function | 4 years
  Change in muscle function assessed by various tests such as:
  6 min walk test: At the 6th minute, the operator also notes the level of dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: MONTASTIER Emilie, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Rangueil Hospital, Toulouse, France, France

IPD SHARING:
Plan to Share IPD: No